CLINICAL TRIAL: NCT01661725
Title: Phase I Clinical Trial of Group ACYW135 Meningococcal Polysaccharide Vaccine
Brief Title: Clinical Trial of Group ACYW135 Meningococcal Polysaccharide Vaccine 001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hualan Biological Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hualanbio-Meningococcal CT 001; Hualanbio-phase I CT (Other Grant/Funding Number: Hualan Biological Engineering Inc.)
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Meningitis
Keywords: Group ACYW135 Meningococcal Polysaccharide Vaccine
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group ACYW135 Meningococcal Polysaccharide Vaccine (Experimental): 0.5ml/ vial
  Interventions: Biological: Group ACYW135 Meningococcal Polysaccharide Vaccine

INTERVENTIONS:
Biological: Group ACYW135 Meningococcal Polysaccharide Vaccine — 60 subjects were divided into three groups (20 subjects each group), adult (16~30 years of age), early youth (7~15 years of age) and children (2~6 years of age) to receive Group ACYW135 Meningococcal Polysaccharide Vaccine, 0.5 ml, one dose regime
  Other Names: Hualan Bio

SUMMARY:
The clinical trial was designed to evaluate the safety against Group ACYW135 Meningococcal Polysaccharide Vaccine of Hualan administered on subjects 2 years of age and older.

DETAILED DESCRIPTION:
Complying with requirements of the approval letter of clinical trial issued by SFDA (Approval Letter No.: 2006L01017), Hualan conducted phase I clinical trial of Group ACYW135 Meningococcal Polysaccharide Vaccine. The safety end points were the presence of any systemic, local and adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy permanent residence 2 years of age and older, the subjects (or their guardians) are able to understand and sign the informed consent;
* Healthy male or female by oral history, physical examination and clinical judgment and who complies with vaccination of this product;
* Be able to comply with the requirements of clinical trial protocol and immunogenicity examination;
* Have no history of vaccination within the past 3 months and vaccination with other products within the last 2 weeks;
* Axillary temperature ≤37.0℃.

Exclusion Criteria:

* Any acute disease, such as: tumor, autoimmunity disease, progressive atherosclerotic disease or diabetes with complication, chronic obstructive pulmonary disease need oxygen uptake, acute or progressive hepatopathy or nephropathy, congestive heart-failure, etc.;
* Allergic to vaccines or drugs (history of allergy to any vaccine in the past);
* History of neurologic symptom or signs;
* Known or suspected (or high risk) impaired or abnormal immune function, e.g.: receive immunosuppressant or immunopotentiator therapy, take immunoglobulin or blood product or plasma extract (except the gastrointestinal tract) within the past 3 months, HIV infection or related disease, etc.;
* History of meningitis infection or vaccination of meningococcal vaccine within the past 3 months;
* History of receiving other vaccines or immunoglobulin injection or any research drugs;
* Any acute disease needing application of antibiotics or anti-virus treatment in the whole body within the past 1 week;
* History of fever within the past 3 days (axillary temperature ≥38.0℃);
* Participating in another clinical trial;
* History of allergy, eclampsia, epilepsy, encephalopathy and mental disease or family disease;
* Thrombopenia or other coagulopathy that may cause contraindication to intramuscular injection;
* Acute chronic disease (such as Down syndrome, diabetes, sickle cell anemia or neurologic disease, Guillain-Barre Syndrome);
* Known or suspected diseases, including: respiratory system disease, acute infection or active stage of chronic disease, SBAV infection of children or mothers, cardiovascular disease, acute hypertension, cancer treatment, skin disease, etc.;
* Pregnancy;
* Any condition that, in the judgment of investigator, may affect trial assessment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2006-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety | Day 28 after vaccination
  All systemic and local adverse reactions and related adverse events on day 28 after the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fubao Ma, Bachelor, Principal Investigator — Immunization Program Institute of Jiangsu Provincial Center for Disease Control and Prevention